CLINICAL TRIAL: NCT04846348
Title: An Open-Label Pilot Study to Evaluate the Effectiveness and Tolerability of a Topical Composition Therapy for the Treatment of Cutaneous Mastocytosis
Brief Title: Topical Composition Therapy for the Treatment of Cutaneous Mastocytosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: It was difficult to enroll patients during the pandemic. A new oral drug, Avapritinib, has since been approved for systemic mastocytosis. This medication controls skin manifestations of mastocytosis and is more convenient for patients to use.
Sponsor: Joseph Butterfield (Other)
Responsible Party: Sponsor-Investigator, Joseph Butterfield, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-011876
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Results first posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-03

CONDITIONS: Cutaneous Mastocytoses
MeSH Terms: conditions — Mastocytosis, Cutaneous | interventions — Diphenhydramine; trolamine salicylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Skin Guard (Experimental): Skin cream combination of ingredients includes 2 agents which target mast cell mediators and one agent which globally reduces mast cell degranulation combined in an emollient cream base:
  Vanicream: Over the counter emollient cream Diphenhydramine Antihistamine Trolamine salicylate Prostaglandin inhibitor, antiinflammatory Cromolyn Sodium Mast cell degranulation inhibitor
  Interventions: Combination Product: Topical preparation of sodium cromolyn 5%, diphenhydramine 1% and trolamine salicylate 10% in emollient cream base.

INTERVENTIONS:
Combination Product: Topical preparation of sodium cromolyn 5%, diphenhydramine 1% and trolamine salicylate 10% in emollient cream base. — Combination of ingredients includes 2 agents which target mast cell mediators and one agent which globally reduces mast cell degranulation combined in an emollient cream base (Vanicream).components: Vanicream: Over the counter emollient cream Diphenhydramine Antihistamine Trolamine salicylate Prostaglandin inhibitor, antiinflammatory Cromolyn Sodium Mast cell degranulation inhibitor
  Other Names: Skin Guard

SUMMARY:
The purpose of this study is to determine the effectiveness and tolerability of a novel topical preparation for the treatment of cutaneous lesions of mastocytosis.

ELIGIBILITY:
Inclusion criteria

* Biopsy proven cutaneous mastocytosis with or without evidence of systemic disease
* Male and female patients 18 to 80 years of age
* No UVB treatment of the skin for 6 months prior to study entry
* No use of topical or systemic corticosteroids for 1 month prior to study entry
* Good general health as confirmed by medical history
* Female patients of child-bearing potential with negative urine pregnancy test who agree to use effective methods of birth control or remain abstinent during treatment. Participants must use birth control for the entire study and for at least 1 week after the last application of the study formulation. Acceptable methods of birth control include ongoing hormonal contraception methods, (such as birth control pills, patches, injections, vaginal ring, or implants), barrier methods (such as a condom (for men) or diaphragm used with a spermicide), intrauterine devices, tubal ligation, or abstinence.
* Patients who are willing and capable of cooperating to the extent and degree required by the protocol; and
* Patients who read and sign an approved informed consent for this study

Exclusion criteria

* Vulnerable study population
* Exposure to ultraviolet B (UVB) radiation to any region of the skin surface for 6 months
* Regular use of skin lightening agents within 1 month of study entry, including

  * Topical corticosteroids
  * Topical bleaching products
  * Topical retinoids
* Use of systemic preparations within 1 month of study entry, including:

  * Systemic corticosteroids
  * Systemic cyclosporine, interferon
  * Systemic acitretin, etretinate, isotretinoin
  * Systemic methotrexate,
  * Systemic photoallergic, phototoxic and/or photosensitizing drugs
* UV light therapy and sunbathing
* Inability to communicate or cooperate with the Principal Investigator and/or Investigators due to language problems, poor mental development or impaired cerebral function
* Pregnant or nursing women
* Women planning a pregnancy within the study period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Butterfield, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Skin Guard: Skin cream combination of ingredients includes 2 agents which target mast cell mediators and one agent which globally reduces mast cell degranulation combined in an emollient cream base:
  Vanicream: Over the counter emollient cream Diphenhydramine Antihistamine Trolamine salicylate Prostaglandin inhibitor, antiinflammatory Cromolyn Sodium Mast cell degranulation inhibitor
  Topical preparation of sodium cromolyn 5%, diphenhydramine 1% and trolamine salicylate 10% in emollient cream base.: Combination of ingredients includes 2 agents which target mast cell mediators and one agent which globally reduces mast cell degranulation combined in an emollient cream base (Vanicream).components: Vanicream: Over the counter emollient cream Diphenhydramine Antihistamine Trolamine salicylate Prostaglandin inhibitor, antiinflammatory Cromolyn Sodium Mast cell degranulation inhibitor
Period: Overall Study
Arm/Group | Skin Guard
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Skin Guard
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Cutaneous Symptom Relief
Description: Number of participants who achieve complete resolution or near-complete clearing of cutaneous symptoms of treated, involved skin
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Skin Guard
Number analyzed (Participants) | 1
Participants | 0

2. Primary Outcome: SkinDex-16 Quality of Life Questionnaire
Description: This validated questionnaire is a 16-item, participant-reported survey used to assess quality of life impacts due to the participant's skin condition. Scores range from 0 to 6, where 0 is never bothered by the skin condition and 6 is always bothered by the skin condition. Results are summed to produce an overall score, ranging from 0 to 96, where lower scores indicated a higher level of quality of life.
Time Frame: Baseline
Measure: Number; unit: score on a scale
Arm/Group | Skin Guard
Number analyzed (Participants) | 1
score on a scale | 78

3. Primary Outcome: SkinDex-16 Quality of Life Questionnaire
Description: as for outcome 2
Time Frame: 2 weeks
Measure: Number; unit: score on a scale
Arm/Group | Skin Guard
Number analyzed (Participants) | 1
score on a scale | 75

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant from enrollment until last visit, for approximately two weeks.
Arm/Group | Skin Guard
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
It was difficult to enroll patients during the pandemic. Additionally, a new oral drug, Avapritinib, has since been approved for systemic mastocytosis. This medication controls skin manifestations of mastocytosis and is more convenient for patients to use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT04846348/Prot_SAP_000.pdf